CLINICAL TRIAL: NCT05029050
Title: Alpha 2 Adrenergic Receptor Agonists for the Prevention of Delirium and Cognitive Decline After Open Heart Surgery (ALPHA2PREVENT): Randomised Controlled Trial.
Brief Title: Dexmedetomidine or Clonidine Infusion for Prevention of Delirium After Open Heart Surgery
Acronym: ALPHA2PREVENT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Haukeland University Hospital (Other); University Hospital of North Norway (Other); UMC Utrecht (Other); Sahlgrenska University Hospital (Other); St. Olavs Hospital (Other)
Responsible Party: Principal Investigator, Bjørn Erik Neerland, MD, Medical doctor, postdoctoral researcher, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2021-001645-12; 2021-001645-12 (EudraCT Number)
Record Dates: First submitted 2021-08-21; First posted 2021-08-31 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Delirium; Cognitive Decline; Frailty
Keywords: delirium; cognitive decline; frailty; heart surgery
MeSH Terms: conditions — Delirium; Cognitive Dysfunction; Frailty | interventions — Dexmedetomidine; Clonidine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: A parallel-group treatment, five-centre, participant and investigator masked, three-arm study to assess the safety and effectiveness of dexmedetomidine or clonidine infusion compared to placebo for the prevention of delirium and cognitive decline in male and female participants aged 70+ scheduled for open heart surgery.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dexmedetomidine (D) (Experimental): Continuous intravenous infusion of dexmedetomidine 0.4 μg/kg/hour from the start of cardiopulmonary bypass and during surgery, followed by 0.2 μg/kg/hour until discharge from the ICU or 24 hours postoperatively, whichever happens first.
  Interventions: Drug: Dexmedetomidine
- Clonidine (C) (Experimental): Continuous intravenous infusion of clonidine 0.4 μg/kg/hour from the start of cardiopulmonary bypass and during surgery, followed by 0.2 μg/kg/hour until discharge from the ICU or 24 hours postoperatively, whichever happens first.
  Interventions: Drug: Clonidine
- Placebo (P) (Placebo Comparator): Continuous intravenous infusion of saline 0.4 μg/kg/hour from the start of cardiopulmonary bypass and during surgery, followed by 0.2 μg/kg/hour until discharge from the ICU or 24 hours postoperatively, whichever happens first.
  Interventions: Drug: Natriumchlorid

INTERVENTIONS:
Drug: Dexmedetomidine — Continous intravenous infusion
  Other Names: Dexdor; Precedex; N05C M18
  Arms: Dexmedetomidine (D)
Drug: Clonidine — Continous intravenous infusion
  Other Names: Catapresan; Catapressan; N02C X02
  Arms: Clonidine (C)
Drug: Natriumchlorid — Continous intravenous infusion NaCl
  Other Names: Saline; NaCl 9mg/ml
  Arms: Placebo (P)

SUMMARY:
A parallel-group treatment, five-centre, participant and investigator masked, three-arm study to assess the safety and effectiveness of dexmedetomidine or clonidine infusion compared to placebo for the prevention of delirium and cognitive decline in male and female participants aged 70+ scheduled for open heart surgery.

DETAILED DESCRIPTION:
Delirium is a major public health concern without therapeutic options. It is an acute disturbance of attention and cognition, precipitated by an acute somatic condition. Delirious patients are often subject to off-label treatment with psychotropic drugs that have dubious effects.

The intravenous alpha-2-adrenergic receptor agonist dexmedetomidine, attenuating sympathetic nervous system activity, shows promise as treatment for delirium, but its use is limited to intensive care units (ICU). Its long-term cognitive effects are unknown. Clonidine is a pharmacodynamically similar drug that can be given orally and has been used for decades as an antihypertensive agent, but is else sparsely studied.

ALPHA2PREVENT will be a three-armed randomised controlled trial to study 1) whether repurposing of clonidine can represent a novel treatment option for delirium, and 2) the possible effects of both dexmedetomidine and clonidine on long-term cognitive trajectories, motor activity patterns, patient rated outcome measures and biomarkers of neuronal injury.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

1. Participant must be ≥70 years old at the time of signing the informed consent.
2. Participant must be accepted for cardiac surgery with cardiopulmonary bypass. The surgical procedures may constitute 1) coronary bypass grafting, 2) tricuspid, mitral, or aortic valve replacement or repair, 3) surgery on the ascending aorta, and 4) the combination any of these procedures.
3. Participant must be capable of giving signed informed consent.

   Exclusion Criteria:

   Participants are excluded from the study if any of the following criteria apply:
4. Preoperative delirium
5. Known hypersensitivity to the active ingredient or components of the product
6. Bradycardia due to sick-sinus-syndrome, 2nd or 3rd degree AV-block (if not treated with pacemaker) or any other reason causing HR <50 bpm at time of inclusion
7. Uncontrolled hypotension
8. Ischemic stroke or transitory ischemic attack the last month or critical peripheral ischemia
9. Acute coronary syndrome last 24 hours. Acute coronary syndrome is defined according to international guidelines
10. Left ventricular ejection fraction < 40%
11. Severe renal impairment (estimated GFR <20ml/min) or expected requirement for renal replacement therapy
12. Severe hepatic dysfunction (liver enzyme three times the upper limit of normal together with a serum albumin concentration below the normal reference limit)
13. Reduced peripheral autonomous activity (e.g. spinal cord injury)
14. Current use of tricyclic antidepressants, monoamine reuptake inhibitors or ciclosporin
15. Endocarditis or sepsis
16. Pheochromocytoma
17. Planned deep hypothermia and circulatory arrest
18. Emergency surgery, defined as less than 24 hours from admission to surgery
19. Previously included in this study
20. Not speaking or reading Norwegian
21. Any other condition as evaluated by the treating physician

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2022-01-17 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative delirium | Up to 7 days
  Cumulative incidence of postoperative delirium, as diagnosed according to Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5) criteria

SECONDARY OUTCOMES:
Incidence of coma | Up to 7 days
  Incidence of coma, as measured by Richmond Agitation Sedation Scale (-5 to +5)
Incidence of death, coma or postoperative delirium | Up to 7 days
  Incidence of death, coma or postoperative delirium, as described above
Number of delirium days postoperatively | Up to 7 days
  Number of delirium days postoperatively, as diagnosed according to DSM-5 criteria
Delirium severity | Up to 7 days
  Delirium severity, as measured by Confusion Assessment Method for Intensive Care Units-7 (CAM-ICU)-7
Motor activity patterns | 6 months
  Motor activity patterns, assessed with body worn accelerometers
Change in cognitive function between inclusion and after 1 and 6 months | 6 months
  Change in cognitive function between inclusion and after 1 and 6 months, as graded by Montreal Cognitive Assessment (MoCA), 10-words memory task from The Consortium Establish a Registry for Alzheimer's Disease (CERAD), digit span tests, Trail making tests (TMT) A and B, semantic and phonemic verbal fluency, and measured repeatedly preoperatively and 1 and 6 months after surgery
Change in patient rated health status between inclusion and after 1 and 6 months | 6 months
  Change in patient rated health status between inclusion and after 1 and 6 months, as assessed by the EQ-5D-5L questionnaire preoperatively and 1 and 6 months postoperatively
Serum concentrations of NFL and p-tau181 | 5 days postoperatively
  Comparison to inclusion of serum concentrations of neurofilament light (NFL) and p-tau181 1, 3 and 5 days postoperatively
Estimate associations between frailty and the other endpoints | 6 months
  Estimate associations between frailty and the other endpoints, as described above
Safety and tolerability | 6 months
  Safety and tolerability as determined by the numbers of Adverse Events (AEs), serious AEs (SAEs) and suspected unexpected serious adverse reactions (SUSARs), and vital signs; blood pressure (BP), heart rate (HR), peripheral oxygen saturation (SpO2) postoperatively
Interaction between preoperative frailty and treatment on delirium and the other endpoints | 6 months
  Interaction between preoperative frailty and treatment on delirium and the other endpoints, as described above
Change in frailty status between inclusion and after 1 and 6 months | 6 months
  Change in frailty status between inclusion and after 1 and 6 months, as graded by the frailty index (FI) and essential frailty toolset (EFT) (section 8.1.3), and measured repeatedly preoperatively and 1 and 6 months after surgery
Comparison of change in frailty status between inclusion and after 1 and 6 months | 6 months
  Comparison of change in frailty status between inclusion and after 1 and 6 months (as described above) between patients with or without postoperative delirium.

OTHER OUTCOMES:
Additional biomarkers | 5 days postoperatively
  Additional biomarkers of neural injury, inflammation or neurotransmission may be explored

CONTACTS AND LOCATIONS:
Overall Officials: Bjørn Erik Neerland, PhD, Principal Investigator — Oslo University Hospital
Locations (5):
- Norway (5):
  - Haukeland University Hospital, Bergen
  - Oslo University Hospital Rikshospitalet, Oslo
  - Oslo University Hospital Ullevål, Oslo
  - University Hospital of North Norway, Tromsø
  - St Olav University Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Neerland BE, Busund R, Haaverstad R, Helbostad JL, Landsverk SA, Martinaityte I, Norum HM, Raeder J, Selbaek G, Simpson MR, Skaar E, Skjaervold NK, Skovlund E, Slooter AJ, Svendsen OS, Tonnessen T, Wahba A, Zetterberg H, Wyller TB. Alpha-2-adrenergic receptor agonists for the prevention of delirium and cognitive decline after open heart surgery (ALPHA2PREVENT): protocol for a multicentre randomised controlled trial. BMJ Open. 2022 Jun 20;12(6):e057460. doi: 10.1136/bmjopen-2021-057460. PMID 35725264